CLINICAL TRIAL: NCT05469620
Title: Open-label, Randomized Comparative Clinical Trial on the Clinical Effect of Adaptive Nutrition Therapy in Hemodialysis Patients
Brief Title: Adaptive Nutrition Therapy in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: Hallym University Kangnam Sacred Heart Hospital (Other); KangWon National University Hospital (Other); Korea University Guro Hospital (Other); Korea University Ansan Hospital (Other); Myongji Hospital (Other); Korea Data Agency (Unknown); Eatmapl (Unknown); Daejeon Eulji Medical Center (Unknown); Seoul National University (Other)
Responsible Party: Principal Investigator, Hoseok Koo, Director, Inje University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: DNET_CKD nutrition 1.0
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Renal Dialysis
Keywords: nutrition
MeSH Terms: interventions — Meals; Educational Status

STUDY DESIGN:
Intervention Model Description: 2 by 2 factorial design, consisting of nutrition education and meal kit prescription.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Receive usual care.
- Education (Experimental): Receive nutrition education.
  Interventions: Other: Education
- Meal (Experimental): Receive meal kit.
  Interventions: Dietary Supplement: Meal
- Education and Meal (Experimental): Receive both nutrition education and meal kit.
  Interventions: Dietary Supplement: Meal; Other: Education

INTERVENTIONS:
Dietary Supplement: Meal — Either a meal kit low in sodium, potassium, and phosphorus; or a meal kit low in sodium only is provided based on predefined logic. Meal kits are delivered in bulk twice a week, meant to replace one meal a day.
  Arms: Education and Meal; Meal
Other: Education — Leaflet or video education materials on seven nutrition-related topics are provided, based on predefined logic. Materials are sent throughout the week, via SMS links.
  Arms: Education; Education and Meal

SUMMARY:
8-week adaptive nutrition intervention for participants undergoing hemodialysis, consisting of nutrition education and meal kit.

ELIGIBILITY:
Inclusion Criteria:

* have been on hemodialysis for over 3 months

Exclusion Criteria:

* diagnosed with cancer within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-12-26 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Potassium | 4 weeks
  Serum potassium level measured from routine blood test.
Phosphate | 4 weeks
  Serum phosphate level measured from routine blood test.
Malnutrition | 8 weeks
  10-item nutritional status measured with Malnutrition Inflammation Score. Scores range from 0 to 30, higher value corresponding to worse outcome (higher risk of malnutrition)

SECONDARY OUTCOMES:
Depression | 8 weeks
  21-item depression score measured with Korean-Beck Depression Inventory. Scores rnage from 0 to 63, higher value corresponding to worse outcome (severe depression).
Self-Efficacy | 8 weeks
  10-item Self-Efficacy score for hemodialysis patients. Scores range from 10 to 40, higher values corresponding to better outcome (higher self-efficacy).

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Seoul Paik Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No